CLINICAL TRIAL: NCT03775265
Title: Phase III Randomized Trial of Concurrent Chemoradiotherapy With or Without Atezolizumab in Localized Muscle Invasive Bladder Cancer
Brief Title: Chemoradiotherapy With or Without Atezolizumab in Treating Patients With Localized Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-03264; NCI-2018-03264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1806 (Other: SWOG); S1806 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Bladder Urothelial Carcinoma; Muscle Invasive Bladder Carcinoma; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cystoscopy; Fluorouracil; dehydroftorafur; Gemcitabine; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex; Radiotherapy; Radiation; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (RT, chemotherapy) (Active Comparator): Patients undergo RT (3DCRT or IMRT) daily Monday-Friday for up to 7-8 weeks. Patients also receive chemotherapy based on physician's choice of gemcitabine IV twice weekly for 6 weeks concurrent with RT, or cisplatin IV weekly for 6 weeks concurrent with RT, or fluorouracil IV on same days as doses 1-5 and 16-20 of radiation therapy and mitomycin IV on day 1 of radiation therapy in the absence of disease progression or unacceptable toxicity. Patients also undergo a TURBT with bladder biopsy at randomization and week 18 as well as cystoscopy at randomization, at weeks 18, 30, 42, 54, then every 3 months through year 2, followed by every 6months through year 5 and CT or MRI at randomization, at weeks 18, 30, 42, 54, then every 6 months through year 2, followed by every 12 months through year 5.
  Interventions: Procedure: Biopsy of Bladder; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Cystoscopy; Drug: Fluorouracil; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Other: Survey Administration; Procedure: Transurethral Resection of Bladder Tumor
- Arm II (RT, chemotherapy, atezolizumab) (Experimental): Patients undergo RT (3DCRT or IMRT) daily Monday-Friday for up to 7-8 weeks and receive chemotherapy based on physician's choice as in Arm I. Patients also receive atezolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a TURBT with bladder biopsy at randomization and week 18 as well as cystoscopy at randomization, at weeks 18, 30, 42, 54, then every 3 months through year 2, followed by every 6months through year 5 and CT or MRI at randomization, at weeks 18, 30, 42, 54, then every 6 months through year 2, followed by every 12 months through year 5.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy of Bladder; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Cystoscopy; Drug: Fluorouracil; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Other: Survey Administration; Procedure: Transurethral Resection of Bladder Tumor

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm II (RT, chemotherapy, atezolizumab)
Procedure: Biopsy of Bladder — Undergo a bladder biopsy
  Other Names: Bladder Biopsy
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT or MRI
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Cystoscopy — Undergo a cystoscopy
  Other Names: CS
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Procedure: Magnetic Resonance Imaging — Undergo CT or MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Given IV
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo 3DCRT or IMRT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Other: Survey Administration — Ancillary studies
Procedure: Transurethral Resection of Bladder Tumor — Undergo a TURBT
  Other Names: Transurethral resection (TURBT); TURBT

SUMMARY:
This phase III trial studies how well chemotherapy and radiation therapy work with or without atezolizumab in treating patients with localized muscle invasive bladder cancer. Radiation therapy uses high energy rays to kill tumor cells and shrink tumors. Chemotherapy drugs, such as gemcitabine, cisplatin, fluorouracil and mitomycin-C, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with radiation therapy may kill more tumor cells. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving atezolizumab with radiation therapy and chemotherapy may work better in treating patients with localized muscle invasive bladder cancer compared to radiation therapy and chemotherapy without atezolizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare bladder intact event-free survival (BI-EFS) for concurrent chemoradiation therapy (CRT) with and without atezolizumab in localized muscle invasive bladder cancer (MIBC).

SECONDARY OBJECTIVES:

I. To compare overall survival between the two arms. II. To compare modified bladder intact event-free survival including cancer related death between arms.

III. To compare complete and partial pathologic response between arms at 3 months after completing chemoradiation therapy.

IV. To estimate metastases-free survival by arm. V. To compare the qualitative and quantitative adverse events from each arm. VI. To estimate the rate of non-muscle invasive bladder cancer recurrence by arm.

VII. To estimate the rate of salvage cystectomy and reasons for cystectomy by arm.

VIII. To compare mean patient-reported global quality of life (QOL) at week 54 using the European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30 Global Health Status (GHS) subscale score between patients with localized muscle-invasive bladder cancer randomized to chemoradiation with versus (vs.) without atezolizumab.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To test the hypothesis that a panel of validated biomarkers of concurrent CRT involving nuclear MRE11, impaired deoxyribonucleic acid damage response (DDR) function and tumor subtyping will be prognostic for BI-EFS among patients receiving either concurrent CRT or chemoimmuno-radiotherapy (CIRT) of the primary tumor.

II. To test the hypothesis that tumor total mutation burden, neoantigen burden, infiltrating immune response, PD-L1 expression and T cell response are associated with augmented response after concurrent CIRT.

III. To bank urine specimens for future use.

PATIENT-REPORTED OUTCOMES (PROs) OBJECTIVES:

I. To compare mean patient-reported global QOL as measured by the EORTC QLQ-C30 Global Health Status subscale scores at week 54 between patients with localized muscle-invasive bladder cancer randomized to chemoradiation with vs. without atezolizumab. (Primary) II. To compare mean patient-reported bowel symptoms at each assessment time by arm using the Expanded Prostate Cancer Index Composite (EPIC) Bowel Assessment from the Expanded Prostate Index, the bladder-specific supplement to the QLQ-C30, the EORTC QLQ-Muscle Invasive Bladder Cancer (BLM30), the Physical Functioning subscale of the EORTC QLQ-C30, and overall health status using the EuroQol Five Dimension Five Level Scale (EQ-5D-5L). (Exploratory) III. To compare longitudinal change over time by arm in patient-reported global QOL using the EORTC QLQ-C30, the Bowel Domain of the Expanded Prostate Index (EPIC Bowel Assessment), the bladder-specific supplement to the QLQ-C30, the EORTC QLQ-BLM30, the Physical Functioning subscale of the EORTC QLQ-C30, and overall health status using the EQ-5D-5L. (Exploratory)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo radiation therapy (RT) (3 dimensional [D] CRT or intensity-modulated radiation therapy [IMRT]) daily Monday-Friday for up to 7-8 weeks. Patients also receive chemotherapy based on physician's choice of gemcitabine intravenously (IV) twice weekly for 6 weeks concurrent with RT, or cisplatin IV weekly for 6 weeks concurrent with RT, or fluorouracil IV on same days as doses 1-5 and 16-20 of radiation therapy and mitomycin IV on day 1 of radiation therapy in the absence of disease progression or unacceptable toxicity. Patients also undergo a transurethral resection of bladder tumor (TURBT) at randomization and week 18 as well as cystoscopy at randomization, at weeks 18, 30, 42, 54, then every 3 months through year 2, followed by every 6 months through year 5 and computed tomography (CT) or magnetic resonance imaging (MRI) at randomization, at weeks 18, 30, 42, 54, then every 6 months through year 2, followed by every 12 months through year 5.

ARM II: Patients undergo RT (3DCRT or IMRT) daily Monday-Friday for up to 7-8 weeks and receive chemotherapy based on physician's choice as in Arm I. Patients also receive atezolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a TURBT with bladder biopsy at randomization and week 18 as well as cystoscopy at randomization, at weeks 18, 30, 42, 54, then every 3 months through year 2, followed by every 6 months through year 5 and CT or MRI at randomization, at weeks 18, 30, 42, 54, then every 6 months through year 2, followed by every 12 months through year 5.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION: If this will be the first patient from a registering site to receive a given RT modality (3DCRT vs. IMRT), the site must first submit pre-RT planning documents within 3 days of Step 1 registration and receive approval from Imaging and Radiation Oncology Core (IROC) before randomizing the patient to Step 2. If this will not be the first patient to receive a specific RT modality, the patient should be immediately randomized to Step 2 on the same day.
* STEP 2 RANDOMIZATION: If patient required review of pre-RT planning, randomization must occur within 14 days of initial registration.
* Patients must have histologically proven, T2-T4a N0M0 urothelial carcinoma of the bladder within 120 days prior to randomization and no intervening treatment between the histologic proof and randomization. Patients with mixed urothelial carcinoma will be eligible for the trial, but the presence of small cell carcinoma will make a patient ineligible. Patients with lymph nodes >= 1.0 cm in shortest cross-sectional diameter on imaging (computed tomography [CT]/magnetic resonance imaging [MRI] of abdomen and pelvis) must have a biopsy of the enlarged lymph node showing no tumor involvement within 70 days prior to randomization. These patients may be suitable for neoadjuvant chemotherapy and radical cystectomy and are eligible for this trial if they seek out a bladder sparing treatment strategy, however patients who have received prior systemic chemotherapy for bladder cancer are not eligible for the trial.
* Patients must undergo a transurethral resection of bladder tumor (TURBT) within 70 days prior to randomization. In a situation where a patient is referred from outside to the enrolling institution, patient must have a repeat office cystoscopy by the urologist who will be following the patient on the clinical trial to assess the adequacy of the prior TURBT. This cystoscopy can be performed in urologist office without general anesthesia. Patient may then undergo repeat TURBT if deemed necessary as standard of care by the treating urologist. Patients may have either completely or partially resected tumors as long as the treating urologist attempted maximal resection. Patient must not have T4b disease
* Patients must undergo radiological staging within 70 days prior to randomization. Imaging of chest, abdomen, and pelvis must be performed using CT or MRI. Patients must not have evidence of T4bN1-3 disease. Eligibility is based on the local radiology report.
* Patients with hydronephrosis are eligible if they have unilateral hydronephrosis and kidney function meets criteria specified.
* Patients must not have had urothelial carcinoma or histological variant at any site outside of the urinary bladder within the previous 24 months except Ta/T1/carcinoma in situ (CIS) of the upper urinary tract including renal pelvis and ureter if the patient had undergone complete nephroureterectomy.
* Patients must not have diffuse CIS based on cystoscopy and biopsy.
* Patient must be planning to receive one of the protocol specified chemotherapy regimens.
* All adverse events associated with any prior surgery and intravesical therapy must have resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade =< 2 prior to randomization.
* Patient must not have received any systemic chemotherapy for their bladder cancer.
* Patient must not have had prior pelvic radiation.
* Patients must not have received prior treatment for muscle invasive bladder cancer including neoadjuvant chemotherapy for the current tumor.
* Patients must not have received any systemic therapy (including, but not limited to, interferon alfa-2b, high dose IL-2, pegylated interferon [PEG-IFN], anti-PD-1, anti-PD-L1), for non-muscle invasive bladder cancer. Prior intravesical bacillus Calmette-Guerin (BCG), interferon, and intravesical chemotherapy are allowed.
* Patients must not have received any of the following prohibited therapies within 28 days prior to randomization or be planning to receive any of the following prohibited therapies during protocol treatment:

  * Anti-cancer systemic chemotherapy or biological therapy not specified in the protocol.
  * Immunotherapy not specified in this protocol.
  * Systemic or intravesical use of any non-study anti-cancer agent (investigational or non-investigational).
  * Investigational agents other than atezolizumab.
  * Live vaccines: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines, and are not allowed. Prior administration of intravesical BCG is allowed.
  * Glucocorticoids for any purpose other than to modulate symptoms from an event of suspected immunologic etiology. The use of physiologic doses of corticosteroids (defined as 10 mg prednisone) are acceptable, however site investigators should consult with the study chair for any dose higher than 10 mg prednisone. Dexamethasone 4 mg IV with chemotherapy to prevent nausea is allowed.
  * RANKL infusion: Concurrent denosumab (which binds the cytokine RANKL) for any known indication is prohibited due to interaction with study medication.
* Patients must not have a major surgical procedure within 28 days prior to randomization. If patient had any surgical procedure then they should have recovered to full presurgical performance status and surgical adverse events should have resolved to grade =< 2. TURBT is not considered a major surgical procedure.
* Patients must not have received treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 14 days prior to randomization. Exceptions:

  * Patients may have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea).
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed. Physiological doses equivalent of 10 mg prednisone daily are allowed. Short term steroids given as antiemetic therapy, e.g. 4 mg dexamethasone or equivalent once a week, is allowed.
* Patients must not have received a live, attenuated vaccine within 4 weeks prior to randomization or anticipate that such a live, attenuated vaccine will be required while on protocol treatment and up to 5 months after the last dose of protocol treatment.

  * Inactivated influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to randomization or while on protocol treatment and up to 5 months after the last dose of protocol treatment.
* Patients must not have undergone prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Patients must be >= 18 years of age
* Patient may or may not be radical cystectomy candidates.
* Absolute neutrophil count (ANC) >= 1,500/microliter (mcL) (within 28 days prior to randomization).
* Platelets >= 100,000/mcL (within 28 days prior to randomization).
* Hemoglobin >= 9 g/dL (within 28 days prior to randomization).
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except patients with Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL) (within 28 days prior to randomization).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x IULN (within 28 days prior to randomization).
* Patients must not have clinically significant liver disease that precludes patient from treatment regimens prescribed on the study (including, but not limited to, active viral, alcoholic or other autoimmune hepatitis, cirrhosis or inherited liver disease).
* Patients must have adequate renal function as evidenced by calculated creatinine clearance >= 25 mL/min. The creatinine used to calculate the clearance result must have been obtained within 28 days prior to randomization.
* Patients must have Zubrod performance status =< 2.
* Patients must have a baseline electrocardiography (ECG) performed within 30 days prior to randomization.
* Patient must not have history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis.
* Patients must not have an active infection requiring oral or IV antibiotics within 14 days prior to randomization. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are not eligible. If patient develops urinary tract infection after TURBT they must have recovered from the infection prior to registration.
* Patients must not have active autoimmune disease that has required systemic treatment in past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Autoimmune diseases include, but are not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, Graves' disease treated with methimazole or glomerulonephritis.
* Patient must not have a history of active tuberculosis.
* If patient has a known history of hepatitis B virus (HBV) or hepatitis C virus (HCV), they must meet the following criteria within 28 days prior to randomization.

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
* Patients who are known to be positive for human immunodeficiency virus (HIV) are eligible only if they have all of the following:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests within 28 days prior to randomization.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for two years. Patients with localized prostate cancer who are being followed by an active surveillance program are also eligible.
* Female patients of childbearing potential must have a serum pregnancy test prior to randomization. Patients must not be pregnant or nursing due to the potential teratogenic side effects of the protocol treatment. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of protocol treatment, and for 5 months (150 days) after the last dose of all study drugs. A woman is considered to be of "reproductive potential" if she has had a menses at any time in the preceding 12 consecutive months.
* Patients must not be known to be allergic to Chinese hamster egg or ovary cell products and must not have any known major allergic reactions to any study drug.
* Patients must be offered the opportunity to participate in specimen banking for future studies.
* Patients who can complete Patient-Reported Outcome instruments in English or Spanish must agree to complete the EORTC QLQ-C30, the EORTC QLQ-BLM30, the EPIC Bowel Assessment, and the EQ-5D-5L per protocol schedule of assessment.
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Bladder intact event-free survival (BI-EFS) | From the date of randomization to the first documentation of a BI-EFS event, assessed up to 5 years
  At each time point, futility will be evaluated, and in the latter two analyses, efficacy will also be evaluated as specified. The final BI-EFS intent-to-treat analysis will be conducted using a stratified logrank test stratifying on stratification factors, and testing treatment at the one-sided significance level of 0.022 to account for multiple interim testing. The hazard ratio (HR) will be estimated using a stratified Cox proportional hazards model and the 95% confidence interval (CI) for the HR will be provided. Results from an unstratified analysis will also be provided. Kaplan-Meier methodology will be used to estimate the median BI-EFS for each treatment arm.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to death from any cause, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology for each treatment arm. Will be analyzed using a similar method as for BI-EFS.
Modified bladder intact event-free survival (mBI-EFS) | From date of randomization to the first documentation of a mBI-EFS event, assessed within 90 days
  Analysis of modified BI-EFS, i.e., a sensitivity analysis of BI-EFS, where bladder cancer event is defined as histologically proven presence of muscle invasive bladder cancer, clinical evidence of nodal or metastatic disease, radical cystectomy, or death within 90 days of receiving protocol specified treatment, will also be conducted.
Biopsy response | At 18 weeks
  The Cochran-Mantel-Haenszel statistic will be used with modified ridit scores to evaluate the biopsy outcomes of complete response versus (vs.) down-staging vs. no response for the two treatment arms.
Complete response duration | From the date of the biopsy documenting the complete response to the time of muscle invasive recurrence, local progression, evidence of metastatic disease or death due to any cause, assessed at 18 weeks
  For the subset of patients who achieve a complete response during the week 18 biopsy window, complete response duration is defined from the date of the biopsy documenting the complete response to the time of muscle invasive recurrence, local progression, evidence of metastatic disease or death due to any cause. Will be analyzed using a similar method as for BI-EFS.
Progression-free survival | From date of randomization to first radiologic or histologic evidence of local progression, nodal or distant metastasis, or death due to any cause, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology for each treatment arm. Will be analyzed using a similar method as for BI-EFS.
Metastasis-free survival | From date of randomization to first radiologic or histologic evidence of metastatic disease or death due to any cause, assessed up to 5 years
  Will be estimated using Kaplan-Meier methodology for each treatment arm. Will be analyzed using a similar method as for BI-EFS.
Cancer-specific survival | From date of randomization to date of death due to bladder cancer, assessed up to 5 years
Quality of life | Baseline up to 5 years
  Assessed with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ)-C30. Will be examined using linear mixed models with patient considered as the random effect. The baseline physical function score and the stratification factors will be included in the regression model as adjustment covariates.

OTHER OUTCOMES:
Treatment interactions | Up to 5 years
  A Cox regression model will be used to evaluate the main effects of treatment arm and the main effect for each stratification factor and the interaction of the stratification factor with treatment in terms of both the primary endpoint and secondary endpoints. The stratification factors to be evaluated include: (1) clinical stage T2 vs. T3/T4a, (2) intended chemotherapy regimen cisplatin vs. 5-FU + mitomycin-C vs. gemcitabine, (3) radiation field small pelvis vs. bladder only and (4) performance status 0-1 vs. 2. There may be other radiation summary measures that may also be explored in terms of their modification of the experimental treatment effect including extent of radiation to lymph node fields. Subgroup analysis defined by stratification factors will also be conducted for primary endpoint and key secondary.

CONTACTS AND LOCATIONS:
Overall Officials: Parminder Singh, Principal Investigator — SWOG Cancer Research Network
Locations (366):
- United States (366):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Sarasota Memorial Hospital-Venice, N. Venice, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group - Urology Robotic and Minimally Invasive Surgery, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Center at University Parkway, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Stephens Hospital, Norway, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT03775265/ICF_000.pdf